CLINICAL TRIAL: NCT04773899
Title: L'Étude de la Dysfonction endothéliale Dans la Maladie à COVID-19 Chez Des Patients en Soins Critiques.
Brief Title: COVID-19 Associated Endothelial Dysfunction Study
Acronym: CAUSED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-A00330-41
Record Dates: First submitted 2021-02-19; First posted 2021-02-26 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Covid19; Microcirculation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort C1 (Other): COVID19 (+) ICU patients with COVID19 pneumonia.
  Interventions: Diagnostic Test: Procedure : Multimodal microvascular assessment at study inclusion
- Cohort C2 (Other): COVID19 (-) matched ICU patients
  Interventions: Diagnostic Test: Procedure : Multimodal microvascular assessment at study inclusion
- Cohort C3 (Other): COVID19 (-) ASA 1 non-hospitalized patients
  Interventions: Diagnostic Test: Procedure : Multimodal microvascular assessment at study inclusion

INTERVENTIONS:
Diagnostic Test: Procedure : Multimodal microvascular assessment at study inclusion — * Vascular occlusion test (VOT) performed on the arm. Measurement of the quality of tissue reperfusion by NIRS on the thenar eminence and the digital perfusion index.
  * Microcirculation reactivity is measured for each patient with a laser speckle contrast imaging (LSCI) placed on the forearm. Tests will be performed for evaluation of microvascular reactivity: Acetylcholine and Nitroprusside Iontophoresis.
  * Morphological analysis of the microcirculation by sublingual videomicroscopy.

SUMMARY:
SARS-CoV-2 enters human cells through the binding of the spike protein with angiotensin converting enzyme-2 (ACE2), a membrane receptor highly expressed in immune or non-immune cells, and in many organs, including lungs and endothelial cells.

In COVID-19 disease, the infection of endothelial might cause an acute endothelial dysfunction.

The objective of this study is to demonstrate that patients COVID19 (+) hospitalized in ICU present an acute endothelial dysfunction (compared with COVID19 (-) also hospitalized in ICU).

This acute endothelial dysfunction could lead to organ failure, systemic immune dysregulation and thrombosis.

DETAILED DESCRIPTION:
This cohort study compares 3 exposure cohorts :

Cohort C1 includes COVID19 (+) patients admitted in ICU in whom the diagnosis of COVID19 pneumonia was confirmed.

Cohort C2 includes COVID 19 (-) matched patients also admitted in ICU.

Cohort C3 is a control group. Patients with few comorbidities, ASA 1, recruited during preoperative assessment for elective surgery.

Eligible patients are included within 72 hours of ICU admission (C1, C2) or during the preoperative assessment (C3). Oral consent is needed after complete explanation of the protocol.

During inclusion visit (V0), patient characteristics as treatments, medical history, clinical and biological data are registered.

Microcirculation is assessed for each patient directly after inclusion.

For patients in C1 and C2 a follow-up is planned. This visit (V1) occurs when the patient is discharged from ICU or the day of his death if it occurs in ICU. In case of prolonged stay in ICU, V1 is carried out 2 months after inclusion. During V1, arterial and/or venous thromboembolic events and mortality in ICU is registered.

For Patients in C3, no follow-up is planned.

ELIGIBILITY:
Inclusion criteria :

* Adult patient (≥ 18 ans)
* Affiliation to the French National Healthcare System
* Voluntary patient who have given oral consent

Cohort C1, COVID19 (+) patients hospitalized in ICU :

* Patient admitted to ICU within 72 hours before inclusion
* Patient presenting SARS-COV2 pneumonia diagnosed by CT scan or by COVID-19 PCR test.

Cohort C2, COVID19 (-) patients hospitalized in ICU :

* Patient admitted to ICU within 72 hours before inclusion
* All COVID19 PCR tests carried out in the 15 days prior inclusion are negative
* All the CT scans possibly performed since the acute event do not show COVID19 pulmonary lesions
* Matching with the cases C1 COVID 19 (+) patients on sex, age (threshold at 65 years), treated hypertension, treated diabetes mellitus.

Cohort C3, elective surgery patients who are not hospitalized in ICU :

* ASA 1 classification (no major comorbidity, a normaly healthy patient)
* Asymptomatic to COVID19 according to French Anesthesiology Society 2020 :

  * No major symptoms among : measured fever > 38°C, dry cough, shortness of breath or high respiratory rate (>20/min), anosmia, ageusia
  * No more than one minor symptom among : sore throat, rhinorrhea, chest pain, myalgia, general alteration or severe tiredness, confusion, disorientation, headache, diarrhea, nausea or/and vomiting, rash/ frostbite/cracking on fingers or hand
* No positive COVID19 PCR test within 15 days prior to inclusion

Non-inclusion criteria :

* Proven sepsis (Procalcitonin >1.0 µg/l) in the 24 hours prior to inclusion
* End-stage kidney disease with dialysis
* Patient with haemodynamic failure treated by norepinephrine
* Patient with traumatic brain injury
* Intubated patient and/or sedated
* Pregnant woman, parturient and nursing mother
* Person restricted in liberty by an administrative or judicial decision
* Patient concerned with admission for psychiatric care
* Adult person subject to a legal protection measure or unable to express consent

Exclusion criteria :

• Cohorts C2 and C3 : positive COVID-19 PCR test within 5 days after inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Endothelial function measured by Near-infrared spectroscopy (NIRS) | within 72 hours of admission in Intensive Care Unit (ICU)
  Measure : Saturation Tissue (StO2) after a vascular occlusion test (VOT)

SECONDARY OUTCOMES:
Endothelial function measured by perfusion index | within 72 hours of admission in ICU
  measure : Perfusion index after a vascular occlusion test (VOT)
Microvascular reactivity measured laser speckle contrast imaging | within 72 hours of admission in ICU
  measure : Vasodilation after iontophoresis of Acetylcholine and Nitroprusside
Morphological analysis by Sublingual videomicroscopy | within 72 hours of admission in ICU
  measure : Microvascular flow index (MFI)
Morphological analysis by Sublingual videomicroscopy | within 72 hours of admission in ICU
  measure : Perfused vessel density (PVD)
Inflammatory status | Inclusion
  measure : C-reactive protein level
Inflammatory status | Inclusion
  measure : neutrophil to lymphocyte ratio
Prothrombotic condition | Inclusion
  measure : D-Dimer Level and
Thrombotic events | Inclusion (V0) up to 8 weeks maximum
  measure : All arterial and/or venous thromboembolic events since acute episode
Severity of lung disease | Inclusion
  measure : PaO2/FiO2 ratio
Severity of lung disease | Inclusion
  measure : percentage of pulmonary lesions assessed by CT scan at the ICU admission.
Mortality | Up to 8 weeks after inclusion
  measure : Mortality in ICU
Organ failure | Inclusion
  measure : Sequential Organ Failure Assessment (SOFA) Score, minimum value 0 and maximum value 24. The higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Samir HENNI, MD PhD, Principal Investigator — UH Angers
Locations (2):
- France (2):
  - UH Angers, Angers
  - Hopital E.Herriot - Hospices Civils de Lyon, Lyon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abrard S, Coquet T, Riou J, Rineau E, Hersant J, Vincent A, Cordoval J, Jacquet-Lagreze M, Allaouchiche B, Lukaszewicz AC, Henni S. DETECTION AND QUANTIFICATION OF MICROCIRCULATORY DYSFUNCTION IN SEVERE COVID-19 NOT REQUIRING MECHANICAL VENTILATION: A THREE-ARM COHORT STUDY. Shock. 2024 Nov 1;62(5):673-681. doi: 10.1097/SHK.0000000000002451. Epub 2024 Aug 12. English, French. PMID 39158987